CLINICAL TRIAL: NCT06365346
Title: Dyadic Video-assisted Gamified Group-based Music Breathing Therapy on Enhancing Resilience Among Children With Attention-deficit Hyperactivity Disorder and Their Caregivers: A Pilot Randomized Controlled Trial
Brief Title: Music Breathing Therapy for Children With Attention-deficit Hyperactivity Disorder and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheung Tan, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024.075-T
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Resilience

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dyadic video-assisted gamified group-based music breathing therapy (Experimental): Parent-child dyads in the intervention group will receive video-assisted gamified music breathing therapy comprising 75-minute weekly sessions (first sessions: parents only; reminding 5 sessions: parent-child dyads) delivered face-to-face by a qualified music breathing practitioner with the aid of animations (mainly for sessions involving children) for 6 weeks. The music breathing therapy comprises four breathing phases, namely "Discovery Breathing", "Triangular Breathing", "Silent Breathing", and "Music Breathing".
  Interventions: Behavioral: Dyadic video-assisted gamified group-based music breathing therapy
- Online educational modules (Active Comparator): Parent-child dyads in the control group will receive weekly online educational modules via email for 6 weeks. Such information will include definition, etiology, risk factors, signs and symptoms, and therapeutic interventions (pharmacological and nonpharmacological), its complications, and how to manage it.
  Interventions: Behavioral: Online educational modules

INTERVENTIONS:
Behavioral: Dyadic video-assisted gamified group-based music breathing therapy — Dyadic video-assisted gamified music breathing therapy comprising six 75-min weekly sessions delivered in a group size of 6-8 (first sessions: parents only; reminding 5 sessions: parent-child dyads).
  Arms: Dyadic video-assisted gamified group-based music breathing therapy
Behavioral: Online educational modules — Six weekly educational modules on ADHD and its management via email.
  Arms: Online educational modules

SUMMARY:
This pilot randomized controlled trial aims to evaluate the feasibility (in terms of rates of recruitment, retention, and attendance), acceptability, and potential effects of the dyadic video-assisted gamified music breathing therapy on dyads' resilience, children's emotional and behavioral symptoms, parents' parenting stress, and psychological distress.

DETAILED DESCRIPTION:
Attention-deficit hyperactivity disorder (ADHD) is a prevalent neurodevelopmental disorder characterized by persistent inattention, hyperactivity, and impulsivity that impact various aspects of both the child's and the caregiver's functioning. Evidence shows that cultivating resilience helps children with ADHD manage emotional dysregulation and improve caregivers' psychological well-being. Music breathing therapy - an adaptation of the Bonny Method of Guided Imagery and Music (GIM) - has shown beneficial effects in enhancing resilience and alleviating psychological distress among different populations. However, it remains unclear whether it is a feasible and effective intervention to enhance the resilience of Chinese school-aged children with ADHD and their caregivers.

Aims:

* To determine the feasibility (in terms of rates of recruitment, retention, and attendance), and acceptability of the intervention
* To examine the effects of the dyadic video-assisted gamified music breathing therapy on dyads' resilience, children's emotional and behavioral symptoms, parents' parenting stress, and psychological distress.

Hypotheses:

It is hypothesized that compared with dyads in the control group, those who receive the dyadic video-assisted gamified music breathing therapy will report the following outcomes: higher levels of dyads' resilience, reduced children's emotional and behavioral symptoms, lower levels of parents' parenting stress and psychological distress at immediately post-intervention (i.e., the 6-week follow-up).

ELIGIBILITY:
Inclusion Criteria:

Children

* have a clinically documented diagnosis/suspected ADHD diagnosis according to DSM-5 criteria
* aged 7 to 12 years (school age)
* can read and communicate in Chinese

Parents

* aged 21 years or above
* are the primary caregivers and living together with the child
* can read and communicate in Chinese

Exclusion Criteria:

Children

* have other disabling diseases (physical disability, mental disability, autism) that might limit their full participation in the study.
* have been engaged in any music intervention in the past 6 months

Parents

* are caring for more than one child with a chronic or critical illness or caring for another family member with a chronic illness
* has a diagnosed mental illness, cognitive impairment, or learning problem, and/or is taking regular psychotropic medications that might limit their full participation in the study
* have been engaged in any music intervention in the past 6 months

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Resilience levels of children | Change from baseline assessment to immediate post-intervention
  The Chinese version of Resilience Scale for Children-10 (RS10) will be used to assess participants' levels of resilience. This scale consists of 10 items. rated on a 4-point Likert scale (from 1 to 4). A higher total score indicates higher level of resilience.
Resilience levels of parents | Change from baseline assessment to immediate post-intervention
  The Chinese version of the Connor-Davidson Resilience Scale will be used to assess the caregivers' levels of resilience. This scale consists of 25 items, rated on a 5-point Likert scale from 0 (not true at all) to 4 (true nearly all of the time). A higher total score indicates higher level of resilience.

SECONDARY OUTCOMES:
Children's emotional and behavioral symptoms | Change from baseline assessment to immediate post-intervention
  The Strengths and Difficulties Questionnaire will be used to assess children's emotional and behavioral symptoms in five domains: (1) emotional symptoms, (2) conduct problems, (3) hyperactivity/inattention, (4) peer relationship problems, and (5) prosocial behavior. This scale consists of 25 items, rated on a 3-point Likert scale. A higher total score indicates greater symptom severity for the emotional and behavioral problem domains and greater prosocial behavior for the prosocial behavior domain.
Parenting stress | Change from baseline assessment to immediate post-intervention
  The Parenting Stress Index-Short Form will be used to assess parenting stress across three domains: (1) parental distress, (2) parent-child dysfunctional interaction, and (3) difficult child behavior. The scale consists of 36 items, rated on a 5-point Likert scale. A higher score indicates higher levels of parenting stress.
Parents' psychological distress (i.e., depression, anxiety and stress) | Change from baseline assessment to immediate post-intervention
  The Chinese version of the 21-item Depression Anxiety Stress Scale (DASS-21) will be used to measure caregivers' mental health states of depression, anxiety and stress over the past week. The scale consists of 21 items, rated on a 4-point Likert scale from 0 (did not apply at all over the last week) to 3 (applied very much or most of the time). A higher score indicates higher levels of depression, anxiety and/or stress.
Feasibility outcomes - recruitment rate | Change from baseline assessment to immediate post-intervention
  Recruitment rates will be calculated as the number of participants who consented to participate in the study divided by the number of participants who meet the inclusion criteria.
Feasibility outcomes - retention rate | Change from baseline assessment to immediate post-intervention
  Retention rate will be calculated as the number of participants who have completed the study divided by the number of randomised participants.
Feasibility outcomes - attendance | Change from baseline assessment to immediate post-intervention
  Attendance rates will be calculated as the number of dyads who have completed the sessions
Acceptability of the intervention - level of satisfaction | Immediate post-intervention
  Dyads' perceived satisfaction of the intervention will be assessed using an 12-item investigator-designed satisfaction survey, a higher total score indicates a higher level of satisfaction.
Acceptability of the intervention | Immediate post-intervention
  Semi-structured individual interviews will be used to evaluate the acceptability of the interventuon by exploring dyads' perceptions and experiences of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ankie Tan Cheung, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No